CLINICAL TRIAL: NCT01347788
Title: Dose-Finding Pilot Study of XL184 in Men With Castrate-Resistant Prostate Cancer and Bone Metastases
Brief Title: Cabozantinib (XL184) in Men With Castrate-Resistant Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Matthew R. Smith, MD, PhD, Professor of Medicine, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-005
Record Dates: First submitted 2011-04-11; First posted 2011-05-04 (Estimated); Results first posted 2015-11-17 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-10

CONDITIONS: Prostate Adenocarcinoma
Keywords: Prostate cancer; Castration Resistant; Bone Metastases
MeSH Terms: conditions — Prostatic Neoplasms | interventions — cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1 (Experimental): Dose level 0: cabozantinib 40 mg daily
  Interventions: Drug: cabozantinib
- Cohort 2 (Experimental): Dose level -1: cabozantinib 20 mg daily
  Interventions: Drug: cabozantinib
- Expansion cohort (Experimental): Dose level 0: cabozantinib 40 mg daily
  Interventions: Drug: cabozantinib

INTERVENTIONS:
Drug: cabozantinib — Cabozantinib PO QD
  Other Names: XL84

SUMMARY:
Cabozantinib (XL184) is a new drug that is being developed to treat cancer. Cabozantinib works by blocking the "angiogenesis," or the growth of new blood vessels, to the tumor. This is similar to how several other cancer drugs work but in addition Cabozantinib also blocks other pathways that may be responsible for allowing cancer cells to become resistant to these other "anti-angiogenic" treatments. So far cabozantinib has been investigated in treating brain cancer and a rare form of thyroid cancer. This study will explore lower doses of cabozantinib with the goal to find the most effective, safe, and tolerable dose without undesirable side effects.

DETAILED DESCRIPTION:
Cabozantinib will be taken by mouth daily. The first five treatment cycles will be 21 days. All cycles after that will be 42 days long. Patients will keep a diary to record study drug dosing.

During the screening phase patients will receive a physical exam, blood and urine tests, a bone scan, a CT of the abdomen and pelvis, and an MRI scan of total body. On Day 1 of each cycle patients will receive a physical exam and blood and urine tests. Bone scan, CT and MRI scans will be performed at the start of cycles 3 and 5, and then repeated once every 12 weeks.

Patients will continue to receive study treatment as long as they are receiving benefit from the treatment, do not experience any severe or unmanageable side effects, and disease does not get any worse.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed prostate adenocarcinoma
* Bone metastases confirmed by bone scan
* Current androgen deprivation therapy
* Castration-resistant disease based on progression in bone and/or PSA progression
* Recovered from toxicities related to prior treatment, except alopecia, lymphopenia, other non-clinically significant adverse events
* Life expectancy of greater than 3 months
* Normal organ and marrow function
* Capable of understanding and complying with the protocol requirements
* Agree to use medically accepted methods of contraception
* Able to swallow capsules

Exclusion Criteria:

* More than two prior chemotherapy regimens for metastatic prostate cancer
* Known untreated, symptomatic or uncontrolled brain metastases
* Serious or unhealed wound
* Treatment with anticoagulants
* Previously identified allergy or hypersensitivity to components of the study treatment formulation
* History of a different malignancy unless disease-free for at least 5 years, or basal or squamous cell carcinoma of the skin
* Current antiretroviral therapy
* Uncontrolled hypertension
* Uncontrolled intercurrent illness

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2011-04; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew R Smith, M.D., Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lee RJ, Saylor PJ, Michaelson MD, Rothenberg SM, Smas ME, Miyamoto DT, Gurski CA, Xie W, Maheswaran S, Haber DA, Goldin JG, Smith MR. A dose-ranging study of cabozantinib in men with castration-resistant prostate cancer and bone metastases. Clin Cancer Res. 2013 Jun 1;19(11):3088-94. doi: 10.1158/1078-0432.CCR-13-0319. Epub 2013 Apr 3. PMID 23553848

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 0; Expansion Cohort: Cabozantinib 40 mg daily
- Dose Level -1: Cabozantinib 20 mg daily
Period: Overall Study
Arm/Group | Dose Level 0 | Dose Level -1 | Expansion Cohort
Started | 11 | 10 | 13
Completed | 11 | 10 | 13
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: See Lee et al CCR 2013
Groups:
- Cabozantinib: Final results have been published Clin Cancer Res. 2013 Jun 1;19(11):3088-94. doi: 10.1158/1078-0432.CCR-13-0319. Epub 2013 Apr 3.
  A dose-ranging study of cabozantinib in men with castration-resistant prostate cancer and bone metastases.
  Lee RJ, Saylor PJ, Michaelson MD, Rothenberg SM, Smas ME, Miyamoto DT, Gurski CA, Xie W, Maheswaran S, Haber DA, Goldin JG, Smith MR.
  Author information Massachusetts General Hospital Cancer Center, Boston, Massachusetts 02114, USA. rjlee@partners.org
Arm/Group | Cabozantinib
Number analyzed (Participants) | 34
Age, Continuous [Median (Full Range); unit: years] | 66 [48 to 83]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 34
Region of Enrollment [Number; unit: participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Partial Response in Bone Scan From Baseline to Week 6
Description: Bone scans will be centrally reviewed and categorized based on comparison of week 6 and baseline imaging. Partial response is defined as 30% or greater decrease in bone scan lesion area from baseline to week 6. An adaptive response design to determine the lowest effective cabozantinib dose among three dose levels (dose level +1, dose level 0 and dose level +1) will be employed.
Time Frame: Baseline and Week 6
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2 | Expansion Cohort
Number analyzed (Participants) | 11 | 10 | 13
participants | 9 | 1 | 6

ADVERSE EVENTS:
Time Frame: Over the entire study period
Groups:
- Cohort 3: Dose level 0: cabozantinib 40 mg daily
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Serious Adverse Events (participants affected / at risk) | 1/11 | 0/10 | 1/13
Other Adverse Events (participants affected / at risk) | 2/11 | 0/10 | 2/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=11) | Cohort 2 (N=10) | Cohort 3 (N=13)
venous thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=11) | Cohort 2 (N=10) | Cohort 3 (N=13)
weight loss (General disorders) | 2 (2) | 0 (0) | 2 (2) — resulted in treatment discontinuation in 3 subjects

LIMITATIONS AND CAVEATS:
Lee RJ, Saylor PJ, Michaelson MD, Rothenberg SM, Smas ME, Miyamoto DT, Gurski CA, Xie W, Maheswaran S, Haber DA, Goldin JG, Smith MR. Clin Cancer Res. 2013 Jun 1;19(11):3088-94. doi: 10.1158/1078-0432.CCR-13-0319. Epub 2013 Apr 3.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No